CLINICAL TRIAL: NCT04845048
Title: Active Pharmacovigilance Study of Post-vaccine Adverse Events of Sinovac's/ Butantan Institute Adsorbed COVID-19 (Inactivated) Vaccine
Brief Title: Active Pharmacovigilance Study of Adsorbed COVID-19 (Inactivated) Vaccine
Status: Completed | Type: Observational
Sponsor: Butantan Institute (Other Government)
Responsible Party: Sponsor
Other Study IDs: CFV-01-IB; Instituto Butantan (Other: Fundação Butantan)
Record Dates: First submitted 2021-04-12; First posted 2021-04-14 (Actual); Last update posted 2023-05-22 (Actual); Status verified 2023-05

CONDITIONS: SARS-CoV-2 Acute Respiratory Disease
Keywords: COVID-19; Adsorbed COVID-19 vaccine (inactivated); Pharmacovigilance
MeSH Terms: conditions — COVID-19 | interventions — Vaccines

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Health care professionals between 18 and 59 years old: Health care professionals
  Interventions: Biological: Adsorbed COVID-19 (Inactivated) Vaccine
- General population 75 years old or more: Elderly 75y plus
  Interventions: Biological: Adsorbed COVID-19 (Inactivated) Vaccine
- General population 60 and 74 years old: Elderly between 60-74y
  Interventions: Biological: Adsorbed COVID-19 (Inactivated) Vaccine

INTERVENTIONS:
Biological: Adsorbed COVID-19 (Inactivated) Vaccine — Adsorbed COVID-19 (inactivated) Vaccine manufactured by Sinovac/Butantan Institute

SUMMARY:
This is a prospective cohort study, observational, multicentre, single-arm, post-registration to assess the safety of the Adsorbed COVID-19 (Inactivated) Vaccine Sinovac / Institute Butantan.

DETAILED DESCRIPTION:
. This is a prospective cohort study, observational, multicentre, single-arm, post-registration to assess the safety of the Adsorbed COVID-19 (Inactivated) Vaccine Sinovac / Institute Butantan.

* The immunization schedule is two doses intramuscular injections (deltoid) with a 14-28 days interval.
* There will be 900 participants (300 health care professionals between 18 and 59 years old); 300 participants 75 years old or more; 300 participants between 60 and 74 years old. All participants must be allowed to receive the Adsorbed COVID-19 (inactivated) Vaccine according to the Brazilian Immunization National Plan.
* For safety analysis , the incidence of adverse events after receiving the Adsorbed COVID-19 (inactivated) Vaccine that needed health assistance until 42 days after two-doses immunization schedule.
* The total period of participation in the study will be approximately 60 days after completing the two-dose schedule of the vaccine.
* Active pharmacovigilance studies are essential to assess the safety profile of the vaccine in subgroups that will be included as target populations in the Immunization Program.

ELIGIBILITY:
Inclusion Criteria:

* Adult allowed to receive the Adsorbed COVID-19 (inactivated) Vaccine according to the Immunization National Plan.
* Informed consent form signed by participant.
* Show voluntary intention to participate in the study and availability throughout the study.

Exclusion Criteria:

* History of severe allergic reactions or anaphylaxis to previous vaccines or allergy to any components of the study vaccine.
* History of fever (axillar temperature ≥ 37,8º C) 72 hours before the vaccine
* Be unavailable during the study period.
* Any other condition that, in the opinion of the principal investigator or his/her representative physician, could put the safety/rights of potential participants at risk or prevent them from complying with this protocol.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The population groups included in this study are the categories that have indication of immunization, defined by the national vaccination plan for COVID-19: health care professionals between 18 and 59 years old and elderly participants 60 aged or over
Sampling Method: Non-Probability Sample
Enrollment: 2549 (Actual)
Dates: Start 2021-05-10 (Actual); Primary Completion 2023-03-12 (Actual); Study Completion 2023-03-13 (Actual)

PRIMARY OUTCOMES:
Safety of the Adsorbed COVID-19 (inactivated) Vaccine through the incidence of adverse reactions. | 7 days after each dose of the vaccine
  Frequency of solicited and non-solicited local and systemic adverse reactions according to age group and severity.
Safety of the Adsorbed COVID-19 (inactivated) Vaccine through the incidence of participants who presented adverse reactions according to the age group | 7 days after each dose of the vaccine
  Frequency of participants who presented any solicited and non-solicited local and systemic adverse reactions according to age group and severity.

SECONDARY OUTCOMES:
Safety of the Adsorbed COVID-19 (inactivated) Vaccine through the incidence of adverse reactions which needed medical care in participants >= 18 years. | 42 days after any dose of the vaccine
  Frequency of solicited and non-solicited local and systemic adverse reactions, which required medical care according to the dose and severity.
Safety of the Adsorbed COVID-19 (inactivated) Vaccine through the incidence of adverse reactions which required medical care in participants < 18 years. | 365 days after the second dose of the vaccine.
  Frequency of solicited and non-solicited local and systemic adverse reactions, which required medical care according to the dose and severity.
Safety of the Adsorbed COVID-19 (inactivated) Vaccine through the incidence of adverse reactions. | First 30 minutes after each dose of the vaccine.
  Frequency of solicited and non-solicited local and systemic adverse reactions according to the dose, severity and age group.
Incidence of serious adverse event (AE) | The whole period of study (365 days after the second dose)
  Incidence of serious adverse event
Description of medications used after adverse event (AE) | The whole period of study (365 days after the second dose)
  Description of medications and duration used after adverse event
Incidence of adverse event of special interest (AESI) | The whole period of study (365 days after the second dose)
  Incidence of adverse event of special interest
Incidence of serious adverse event if a subject get pregnant (SAE) | From the recrod of pregnancy until the end of the study or upto the birth.
  Incidence of serious adverse event if a subject get pregnant after received any dose of the vaccine

CONTACTS AND LOCATIONS:
Overall Officials: Marta H Lopes, MD, Principal Investigator — University of Sao Paulo
Locations (3):
- Brazil (3):
  - Centro de Saúde Escola da Faculdade de Medicina de Botucatu - Unesp., Botucatu, São Paulo
  - Centro de Saúde Escola da Faculdade de Medicina de Ribeirão Preto da Universidade de São Paulo (HCFMRP-USP) Dr. Joel Domingos Machado., Ribeirão Preto, São Paulo
  - Centro de Referência de Imunobiológicos Especiais. Hospital das Clínicas da Faculdade de Medicina da Universidade de São Paulo (CRIEHCFMUSP), São Paulo

IPD SHARING:
Plan to Share IPD: Undecided